CLINICAL TRIAL: NCT00013715
Title: Ozone and Rhinovirus-Induced Disease in Asthmatics
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 9004-CP-001
Record Dates: First submitted 2001-03-28; First posted 2001-03-30 (Estimated); Last update posted 2008-08-11 (Estimated); Status verified 2008-08

CONDITIONS: Asthma
Keywords: Asthma; Rhinovirus; Ozone
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
In the U.S., morbidity associated with human rhinovirus (RV) infection represents a major health problem. In asthmatics, up to 80% of asthma exacerbations are associated with upper respiratory infections. Despite evidence that environmental oxidant pollutants, such as ozone, may increase the severity of viral disease, the mechanisms underlying such an effect have not been identified. This study will test the hypothesis that exposure of allergic asthmatic subjects to ambient levels of ozone directly enhances viral disease by increasing infectivity and intensifying virus-induced inflammation.

DETAILED DESCRIPTION:
In mild asthmatics, the study will investigate: (1) if exposure to ozone will enhance the viral infective process in the nasal epithelium, (2) the effect of ozone exposure on RV-induced inflammatory gene expression, mediator release and inflammatory cell influx into the upper and lower airways, and (3) the interactive effects of ozone and RV on airway reactivity. This information will improve our understanding of the risk associated with oxidant pollutant exposure in this population of individuals in whom RV infection may represent a significant health concern.

ELIGIBILITY:
Subjects recruited will be non-asthmatic controls or mild allergic asthmatics using beta-agonists, mostly on an "as needed" basis. Selection criteria will include good general health by medical history and physical examination, no history of smoking, and the absence of respiratory infection in the preceding 6 week period. Subjects will undergo serologic testing and must have a negative test for neutralizing antibodies to RV16 to participate in all but one study of the project.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 1999-09; Study Completion 2003-08

CONTACTS AND LOCATIONS:
Locations (1):
- The Johns Hopkins School of Hygiene and Public Health, Baltimore, Maryland, United States